CLINICAL TRIAL: NCT02993718
Title: Comparison of the Upper Airway Patency by Dexmedetomidine and Propofol Used for Sedation
Brief Title: Sedation by Dexmedetomidine and Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Principal investigator, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WatchPAT
Record Dates: First submitted 2016-12-11; First posted 2016-12-15 (Estimated); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Anesthesia, Spinal
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Intraoperative sedation is performed by using dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- Propofol (Experimental): Intraoperative sedation is performed by using propofol
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — As a loading dose, 0.5 μg/kg dexmedetomidine was administered over 10 min, which was then administered continuously at a dose of 0.2-0.8 μg/kg/h. Sedation was maintained at modified observer's assessment of alertness/sedation scale 3
  Arms: Dexmedetomidine
Drug: Propofol — Propofol was infused continuously via a target-controlled infusion device, and the effect-site concentration was maintained with a range of 0.5-2.0 μg/ml. Sedation was maintained at modified observer's assessment of alertness/sedation scale 3
  Arms: Propofol

SUMMARY:
Under the hypothesis that dexmedetomidine sedation would result in less upper airway obstruction, we evaluated the occurrence of upper airway collapse or the requirement of airway intervention in patients with obstructive sleep apnea during dexmedetomidine or propofol sedation.

ELIGIBILITY:
Inclusion Criteria:

* Surgery under spinal anesthesia
* Intraoperative sedation
* American Society of Anesthesiology physical status 1 or 2
* Apnea/hypopnea index 5-14/h in Watch-PAT 200 analysis

Exclusion Criteria:

* Anatomical defects on upper respiratory tract
* Psychotic disorder
* Drug addition
* Alcohol addition
* body mass index ≥ 35 kg/m2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The occurrence of upper airway obstruction | During the sedation period, an average of 3 hours.
  When end-tidal carbon dioxide was not detected in spite of the respiratory effort during the sedation period, the case will be regarded as the occurrence of upper airway obstruction.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin HJ, Kim EY, Hwang JW, Do SH, Na HS. Comparison of upper airway patency in patients with mild obstructive sleep apnea during dexmedetomidine or propofol sedation: a prospective, randomized, controlled trial. BMC Anesthesiol. 2018 Sep 5;18(1):120. doi: 10.1186/s12871-018-0586-5. PMID 30185146